CLINICAL TRIAL: NCT04665245
Title: Contact Network Transmission Modeling of Healthcare Associated Infections: Symptom-Based Markers for COVID-19 Transmission
Brief Title: Symptom-Based Markers for COVID-19 Transmission
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Alberto Maria Segre, Professor, Chair, Department of Computer Science, University of Iowa
Other Study IDs: 202007450
Record Dates: First submitted 2020-12-10; First posted 2020-12-11 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Positive Patients: The study only includes one cohort: COVID-19 positive patients. Enrollees will not receive any therapeutic intervention; participants will simply report their temperature and any symptoms experienced twice per day for 10 days.

SUMMARY:
In this study, COVID-19 positive patients will be added to a bidirectional texting program to receive daily surveys about their symptoms with the infection. This data will further the understanding of COVID-19 symptom development throughout the infection period, as well as how those symptoms vary at different points of the day. This study will be a single cohort, observational study of COVID-19 patients.

DETAILED DESCRIPTION:
One important approach for decreasing COVID-19 transmission in healthcare settings is to prevent healthcare professionals from working while ill. Currently, facilities are asking screening questions and measuring temperatures to help identify symptomatic healthcare professionals and exclude them from providing patient care. Simulations can be used to inform the effectiveness of different screening approaches, but the results of these simulations depend upon the effectiveness of the intervention, e.g., the ability to identify healthcare professionals on their way to work, or to study the impact of healthcare professionals returning to work too early. Thus, simulations must necessarily depend upon realistic disease parameters: for example, it is suspected that a non-trivial proportion of patients with COVID-19 may be asymptomatic or have minimal symptoms, but the relative size of the asymptomatic subpopulation is unknown.

The plan for this study is to develop a method for granular measurement of twice-daily symptoms from healthcare professionals and other research subjects of similar ages. After being diagnosed, the goal is to determine what symptoms participants have and how long they have had them. This will be done using a previously-developed bidirectional texting platform to query participants about symptoms at least twice a day for ten days post diagnosis. Participants will be asked about subjective symptoms, including fevers, chills, cough, shortness of breath, fatigue, gastrointestinal symptoms, etc. They will also take their temperature twice daily during the recovery period, which will help determine the effectiveness of screening based on symptoms and/or thermometer readings.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Tested positive for COVID-19

Exclusion Criteria:

* Prisoners
* Unable to provide own informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients at the University of Iowa Hospitals & Clinics (UIHC). Approximately 5,000 people have already tested positive for COVID-19 in Johnson County alone, and numbers are continuing to increase. The University of Iowa Hospitals & Clinics see many patients from outside of Johnson County as well.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto M Segre, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COVID-19 Positive Patients
Started | 214
Completed | 196
Not Completed | 18
Not completed — Lost to Follow-up | 18

BASELINE CHARACTERISTICS:
Arm/Group | COVID-19 Positive Patients
Number analyzed (Participants) | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 6 participants did not complete the baseline survey to report their sex.
  Participants
    number analyzed (Participants) | 208
    Female | 128
    Male | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 6 participants did not complete the baseline survey to report their ethnicity.
  Participants
    number analyzed (Participants) | 208
    Hispanic or Latino | 12
    Not Hispanic or Latino | 194
    Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 6 participants did not complete the baseline survey to report their race.
  Participants
    number analyzed (Participants) | 208
    American Indian or Alaska Native | 4
    Asian | 4
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 7
    White | 192
    More than one race | 0
    Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 214

OUTCOME MEASURES:

1. Primary Outcome: Body Temperature
Description: Body temperature taken each morning and evening throughout COVID-19 infection period.
Time Frame: 10 days
Measure: Median (Standard Deviation); unit: degrees Fahrenheit
Units Other Than Participants: Submitted Temperatures
Arm/Group | COVID-19 Positive Patients
Number analyzed (Participants) | 196
Number analyzed (Submitted Temperatures) | 3,827
degrees Fahrenheit
  number analyzed (Submitted Temperatures) | 3827
  (all) | 98.1 (0.85)

2. Primary Outcome: COVID-19 Symptoms
Description: Any symptoms experienced throughout COVID-19 infection period (aches, cough, decreased sense of taste and/or smell, diarrhea, difficulty breathing, headache, nausea, runny nose, sore throat, shortness of breath).
Time Frame: 10 days
Measure: Count of Units; unit: Submitted Symptoms
Units Other Than Participants: Submitted Symptoms
Arm/Group | COVID-19 Positive Patients
Number analyzed (Participants) | 196
Number analyzed (Submitted Symptoms) | 8910
Submitted Symptoms
  Body or muscle aches | 956
  Cough | 1532
  Decreased sense of taste and/or smell | 1669
  Diarrhea | 305
  Difficulty breathing | 141
  Headache | 1140
  Nausea/vomiting | 168
  Runny nose | 1096
  Shortness of breath | 388
  Sore throat | 747
  None | 768

ADVERSE EVENTS:
Time Frame: 10 days.
Arm/Group | COVID-19 Positive Patients
All-Cause Mortality (participants affected / at risk) | 0/214
Serious Adverse Events (participants affected / at risk) | 0/214
Other Adverse Events (participants affected / at risk) | 0/214

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT04665245/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT04665245/ICF_001.pdf